CLINICAL TRIAL: NCT04939129
Title: The Relationship Between The Change in Systolic Blood Pressure and The Pleth Variability Index (PVI) After The Lung Recruitment Maneuver (LRM) to Evaluate Fluid Responsiveness in Open Abdominal Surgeries
Brief Title: Evaluation of Fluid Responsiveness With Pulse Variation Index and Systolic Blood Pressure Changes After Lung Recruitment Maneuver
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-21-468
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-06

CONDITIONS: Pleth Variability Index; Lung Recruitment Maneuver; Fluid Responsiveness
Keywords: pleth variability index; lung recruitment maneuver; fluid responsiveness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The research is terminated by calculating the percentage of PVI changes with SAB formed by LRM after fluid challenge. — Measurements will begin after a hemodynamically stable period in the supine position.Heart rate, central venous pressure, systolic, diastolic and mean arterial pressure, peripheral oxygen saturation, PVI and BIS baseline values (baseline 1) will be recorded.LRM will be automatically adjusted in the mechanical ventilator(30 cm H2O/30 seconds) and all hemodynamic parameters where the maximum change at the end of 30 seconds, will be recorded(after LRM), and the differences initial baseline values will be calculated and recorded as percentages.After the recording of the second values, the crystalloid infusion at 10ml/kg will be made to the patient through the peripheral venous line within 15minutes, new baseline values will be taken before the test(baseline 2).After fluid replacement, LRM will be repeated in the same way. The values after LRM(Fluid Challenge-FC) will be recorded and differences between basal 2 values will be calculated and recorded as percentages.

SUMMARY:
Evaluation of Fluid Responsiveness With Pulse Variation Index and Systolic Blood Pressure Changes After Lung Recruitment Maneuver

DETAILED DESCRIPTION:
After obtaining ethics committee approval, at least 84 patients who will undergo elective open abdominal surgery under general anesthesia in the operating room of the Ministry of Health Ankara City Hospital will be included in the study. The study is a single center, prospective, observational study.

Weight, height, age, gender, BMI (body mass index), ASA information of the patients will be recorded. Induction and anesthesia management will be applied in accordance with the standard working order of the anesthesia clinic. After the patient is taken to the operating table, non-invasive arterial blood pressure monitoring (noninvasive), 5-lead ECG and pulse oximetry, in addition to standard hemodynamic monitoring, Bispectral Index (BIS), temperature and Massimo ® pulse oximeter (Masimo Corp., Irvine, CA, USA). ) will be monitored. General anesthesia induction will be performed with 0.02 mg / kg midazolam, 1mg / kg lidocaine, 1mcg / kg fentanyl and 2mg / kg propofol after preoxygenation in accordance with the routine practice of the anesthesia clinic, and endotracheal intubation will be performed with a suitable tube for the patient to be provided with 0.6mg / kg rocuronium. BIS target value range will be determined as 40-60, and anesthesia maintenance will be provided by modifying the volatile anesthetic concentration and remifentanil infusion dose (0.1-1 mcg / kg / min) in accordance with hemodynamic values. Ventilation mode and ventilation parameters; tidal volume (6-8 ml / kg according to ideal body weight), respiratory rate (12-16) and end-tidal CO2 values in the range of 30-40 mmhg, inspiratory / expiratory ratio 1: 2, positive end expiratory pressure (PEEP) 5 cm H2O and FiO2: will be set as 50%. After the Allen test to be performed preoperatively, radial artery catheterization and invasive blood pressure monitoring of the non-dominant hand, a 7 fr three lumen central catheter will be placed into the right internal jugular vein with ultrasound (USG) and central venous pressure (CVP) monitoring will be performed. These applications are routinely performed in patients scheduled for open abdominal surgery in our clinic. Preferably 16G or 18G , 2 peripheral venous lines will be placed and fluid will not be given before fluid replacement. Measurements will begin after the patient preparation is complete, after a hemodynamically stable period (defined as the period in which the mean arterial blood pressure (MAP) change is <10% within 5 minutes), in the supine position, and when the patient is confirmed by a second observer that there is no spontaneous breathing effort. Hemodynamic parameters; heart rate (HR) (beats / minute), central venous pressure (CVP) (mmHg), systolic arterial blood pressure (SAP) (mmHg), diastolic arterial blood pressure (DAP) (mmHg), mean arterial blood pressure (MAP) ) (mmHg), peripheral oxygen saturation (SpO2), PVI and BIS baseline values (baseline 1) will be recorded. The LRM will be automatically adjusted in the mechanical ventilator to be at 30 cm H2O for 30 seconds, and the test will begin, all hemodynamic parameters, especially SAB and PVI, where the maximum change at the end of 30 seconds, will be recorded (after LRM), and the differences initial baseline values will be calculated and recorded as percentages. After the recording of the second values, the crystalloid infusion at 10 ml / kg will be made to the patient through the peripheral venous line within 15 minutes, 10 minutes after the end of the infusion, new baseline values will be taken before the test (baseline 2). After fluid replacement, LRM will be repeated in the same way. The values after LRM (Fluid Challenge-FC) will be recorded and differences between basal 2 values will be calculated and recorded as percentages. Primary measurement parameters are determined as PVI and SAB, and secondary measurement parameters are HR, DAB, OAB, SpO2, CVP and BIS. The research is terminated by calculating the percentage of PVI changes with SAB formed by LRM after fluid challenge.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 to 3 patients, over 18 years of age who will undergo elective open abdominal surgery under general anesthesia

Exclusion Criteria:

* being over 75 years old, pregnant, who are contraindicated to use anesthetic drugs, BMI <18 and BMI> 40, who used inotropes or vasopressor drugs before or during the operation, with preoperative lung disease, with left ventricular ejection fraction less than 30%, with suspected right ventricular dysfunction (due to chronic obstructive pulmonary disease (COPD) or obstructive sleep apnea syndrome (OSAS)), with moderate to severe valvular disease, with hemodynamic instability in the perioperative period, with severe peripheral vascular occlusion, with liver failure, with renal insufficiency, with intracranial hypertension and with pulmonary hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who will undergo elective open abdominal surgery under general anesthesia in our hospital
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation between systolic blood pressure change after LRM and PVI in patients who will undergo elective open abdominal surgery under general anesthesia | first 30 minutes of general anesthesia
  In this study, the presence of a correlation between systolic blood pressure change after LRM and PVI in patients who will undergo elective open abdominal surgery under general anesthesia, the systolic pressure change in LRM is a non-invasive test that can be used to predict fluid responsiveness. We aim to reduce the invasive procedures required for the measurement of cardiac output used in the evaluation and to develop an alternative method to the use of expensive and not always accessible devices required for measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Oya Kılcı, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biais M, Lanchon R, Sesay M, Le Gall L, Pereira B, Futier E, Nouette-Gaulain K. Changes in Stroke Volume Induced by Lung Recruitment Maneuver Predict Fluid Responsiveness in Mechanically Ventilated Patients in the Operating Room. Anesthesiology. 2017 Feb;126(2):260-267. doi: 10.1097/ALN.0000000000001459. PMID 27922547
- [Background] De Broca B, Garnier J, Fischer MO, Archange T, Marc J, Abou-Arab O, Dupont H, Lorne E, Guinot PG. Stroke volume changes induced by a recruitment maneuver predict fluid responsiveness in patients with protective ventilation in the operating theater. Medicine (Baltimore). 2016 Jul;95(28):e4259. doi: 10.1097/MD.0000000000004259. PMID 27428237
- [Result] Hood JA, Wilson RJ. Pleth variability index to predict fluid responsiveness in colorectal surgery. Anesth Analg. 2011 Nov;113(5):1058-63. doi: 10.1213/ANE.0b013e31822c10cd. Epub 2011 Sep 30. PMID 21965349
- [Result] Yu Y, Dong J, Xu Z, Shen H, Zheng J. Pleth variability index-directed fluid management in abdominal surgery under combined general and epidural anesthesia. J Clin Monit Comput. 2015 Feb;29(1):47-52. doi: 10.1007/s10877-014-9567-5. Epub 2014 Feb 21. PMID 24557584